CLINICAL TRIAL: NCT06167954
Title: Safety and Usability of a Robotic Gait Device for Children and Adolescents With Neurological or Neuromuscular Disease in Their Natural Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXP-I-US
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy; Acquired Brain Injury; Spinal Muscular Atrophy
Keywords: cerebral palsy; acquired brain injury; spinal muscular atrophy; robotics; gait; rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries; Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXPLORER (Experimental): 8 sessions with the robotics gait device in their homes and natural environment for all participants
  Interventions: Device: EXPLORER

INTERVENTIONS:
Device: EXPLORER — 8 sessions of use of the device in the home and the community of the participants

SUMMARY:
The goal of this clinical trial is to analyze the usability and safety of the robotic gait device EXPLORER in children with cerebral palsy, acquired brain injury and spinal muscular atrophy.

Participants will use the exoskeletons in their home and the community and variables regarding safety and usability will be measured and recorded.

DETAILED DESCRIPTION:
Neurological and neuromuscular diseases are the main cause of motor disability in children, leading to the inability to stand and walk in many cases. Robotic devices are a useful tool in the rehabilitation of these children, but most of them are designed to be used in the clinical setting. EXPLORER is a robotic device designed to assist gait in children with motor disability in their homes and the community. The aim of this study is to analyze the safety and usability of the EXPLORER in children with cerebral palsy, acquired brain injury and spinal muscular atrophy.

A test phase will be conducted in order to make some final modifications and improve the device. Some participants of the sample will use the device in 1-3 occasions in a controlled environment.

After these modifications, participants will use the final version of the device in 8 different occasions in their homes and the community in order to prove its safety and usability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy, acquired brain injury or spinal muscular atrophy
* Medical authorization for standing, gait training and weight bearing.
* Informed consent signed by legal guardians.
* Maximum user weight of 60 kg.
* Hip width (between greater trochanters) ≤40 cm.
* Length of the thigh (distance from the greater trochanter to the lateral condyle of the tibia) from 21cm to 36cm.
* Tibia leg length (distance from the lateral condyle of the tibia to the lateral malleolus) from 20cm to 35cm.
* Shoe size ≤40 (EU)

Exclusion Criteria:

* Medical contraindications for standing or walking.
* Non-reducible contractures or heterotropic ossifications above the degrees allowed by the device or out of the trajectory imposed by the device
* Spasticity equal to 4 on the Modified Ashworth Scale at the time of use of the device.
* More than 20º of hip and/or knee non-reducible contractures at the time of using the exoskeleton.
* Necessity to walk with more than 5º of hip abduction.
* Impossibility to reach 5º of ankle dorsiflexion with ir without orthoses.
* Lower length dysmetria that cannot be mitigated with a wedge under the foot.
* Skin lesion on parts of the lower extremities that are in contact with the device.
* History of fracture without trauma.
* Presence of other conditions causing exercise intolerance (such as uncontrolled hypertension, coronary artery disease, arrhythmia, congestive heart failure, severe pulmonary disease).
* Conductual disorders that may interfere with the use of the device or their participation in the study, like impulsiveness.
* Allergy to any of the EXPLORER materials: cotton, nylon, polyester, PPS, PEEK or ABS.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | through study completion, along 8 weeks
  occurrence of any serious adverse event to the participant or the caregiver
Falls prevalence | through study completion, along 8 weeks
  Number of falling events occurred from the participant or caregiver
Skin integrity | through study completion, along 8 weeks
  Occurrence of any injury of the skin in the areas of contact and produced by the use of the device
Pain (Visual Analogic Scale) | through study completion, along 8 weeks
  pain measured by the Visual Analogic Scale (VAS) by the participant and the caregiver, scored from 0 to 10, being 0 "no pain" and 10 "unbearable pain"
Spasticity | through study completion, along 8 weeks
  spasticity measured by the Modified Ashworth Scale (MAS), scored from 0 (no spasticity) to 4 (affected part in rigid flexion or extension)
Heart rate | through study completion, along 8 weeks
  measurement of heart rate
Oxygen saturation | through study completion, along 8 weeks
  measurement of Oxygen saturation when medical prescription
Donning and doffing time | through study completion, along 8 weeks
  Time to don and doff the device to each participant
Number of steps | through study completion, along 8 weeks
  Number of steps taken provided by the device
Walking time | through study completion, along 8 weeks
  Walking time provided by the device
Interventions of the investigators | through study completion, along 8 weeks
  The number of times that the investigators have to intervene in the session in order to avoid damage when the device is being used by the caregiver
Participant satisfaction | at the end of the intervention, 8th week
  Satisfaction of the participant (caregiver) with the device measured by the Quebec User Evaluation of Satisfaction with Assistive Technology 2.0. (QUEST 2.0), scored with a Likert type scale from 0 to 5, being 0 the lowest satisfaction and 5 the highest possible satisfaction with the device
Blood pressure | through study completion, along 8 weeks
  measurement of blood pressure

SECONDARY OUTCOMES:
Acceptability | at the end of the intervention, 8th week
  Analysis of the drop-out rate during the study period
Accessibility of the participant | through study completion, along 8 weeks
  Rate of the participants suitable to use the device
Accessibility of the house | through study completion, along 8 weeks
  Rate of the houses suitable to use the device
Accessibility of the exterior spaces | through study completion, along 8 weeks
  Rate of the exterior spaces that are suitable to use the device

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Infantil Universitario Niño Jesús-Servicio de Rehabilitación, Madrid
  - Hospital Universitario Niño Jesús-Servicio de Neuro Ortopedia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid